CLINICAL TRIAL: NCT00108251
Title: Aldosterone Antagonism in Diastolic Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-010-03S
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Congestive Heart Failure; Diastole
Keywords: controlled clinical trial; Diastole; Echocardiography; exercise tolerance; Heart Failure, Congestive; Receptors, Aldosterone
MeSH Terms: conditions — Heart Failure; Heart Murmurs | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): placebo tablet
  Interventions: Drug: Eplerenone
- 2 (Experimental): eplerenone tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eplerenone — aldosterone receptor blocker
  Other Names: Inspra
  Arms: 1
Drug: Placebo — matching placebo
  Arms: 2

SUMMARY:
The primary purpose of this study is to determine whether eplerenone has a beneficial effect on improving exercise ability in patients with diastolic heart failure.

DETAILED DESCRIPTION:
The objectives of this study are: 1) To evaluate the effect of eplerenone, an aldosterone antagonist, on intermediate functional outcomes in patients with DHF (diastolic heart failure); 2) To evaluate the effect of eplerenone, an aldosterone antagonist, on echocardiographic measures of diastolic dysfunction in patients with DHF.

The study is an double-blind, placebo-controlled study evaluating the effects of eplerenone compared to placebo in patients with DHF. A total of 48 patients with DHF will be randomized in a 1:1 ratio to 1) Placebo (n=24) or to 2) Eplerenone (n=24) in a dose of 25 mg a day for the first 2 weeks followed by uptitration to 50 mg a day for 22 weeks. The primary outcome is an improvement in functional capacity, measured by the distance covered in a 6-minute walk test. Secondary Outcomes include : Change echocardiographic measures of diastolic dysfunction, change in levels of B-type natriuretic peptide (BNP)and change in quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have DHF as defined by all 3 of the following criteria:

   i)Presence of clinical heart failure for greater than or equal to 2 months before the screening visit. At the time of enrollment they should have NYHA functional class II or III heart failure symptoms such as dyspnea, fatigue on exertion, paroxysmal nocturnal dyspnea, and orthopnea.

   ii)Left ventricular ejection fraction greater than or equal to 50% (by echo, radionuclide angiography or contrast angiography) within 2 months of screening iii) BNP (brain natriuretic peptide) greater than or equal to 62 pg/ml within 2 months of screening
2. Patients euvolemic on clinical examination. If patients are not euvolemic, all attempts will be made to achieve a euvolemic state with change in diuretic doses prior to enrollment into the study
3. Systolic blood pressure less than or equal to 150 mmHg and diastolic blood pressure less than or equal to 95 mmHg for 4 weeks prior to and at the time of enrollment
4. Able to walk at least 50 m at the time of enrollment
5. All patients will be required to be on ACE inhibitors or angiotensin receptor blockers for at least 4 weeks prior to enrollment

Exclusion Criteria:

1. Patients requiring eplerenone or spironolactone for treatment of other comorbid illnesses, e.g. ascites due to cirrhosis. Also, patients with severe hepatic impairment will not be included.
2. Contraindication to eplerenone therapy with creatinine > 2.5 mg/dl or serum potassium > 5.0 mEq/L or creatinine clearance < 30 ml/min/1.73 m2 or intolerance to eplerenone or spironolactone in the past
3. Significant valvular heart disease, pericardial disease or severe chronic lung disease with cor pulmonale, as the cause of symptoms and signs of CHF
4. Patients with technically inadequate echocardiographic windows or patients with severe mitral annular calcification
5. Unstable angina or MI within 4 weeks prior to enrollment
6. Patient with severe peripheral vascular disease and claudication or other physical conditions that will limit the distance walked by them
7. Pregnant or lactating females
8. History of alcohol or substance abuse or history of repeated non-compliance with medications
9. History of cancer within 3 years (other than resected cutaneous basal or squamous cell carcinoma)
10. Participation in any other drug trial within 30 days prior to enrollment
11. Inability to provide informed consent
12. On drugs that are strong inhibitors of CYP3A4 such as ketoconazole, itraconazole, nefazodone, trolandeomycin, clarithromycin, ritonavir, nelfinavir etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-08; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Change in Six Minute Walk Distance from baseline to 24 weeks after randomization | 24 weeks
  change in six minute walk distance between the placebo and spironolactone group

SECONDARY OUTCOMES:
Change in left ventricular stiffness at 24 weeks, Change in other echocardiographic measures of diastolic dysfunction at 24 weeks, Change in levels of B-type natriuretic peptide (BNP) at 24 weeks; Change in quality of life at 24 weeks | 24 weeks
  change in above echocardiogtraphic measures between placebo and spironolactone group

CONTACTS AND LOCATIONS:
Overall Officials: Anita Deswal, MD MPH MBBS, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (1):
- Michael E DeBakey VA Medical Center, Houston, Texas, United States

REFERENCES:
- [Result] Deswal A, Richardson P, Bozkurt B, Mann DL. Results of the Randomized Aldosterone Antagonism in Heart Failure with Preserved Ejection Fraction trial (RAAM-PEF). J Card Fail. 2011 Aug;17(8):634-42. doi: 10.1016/j.cardfail.2011.04.007. Epub 2011 May 31. PMID 21807324